CLINICAL TRIAL: NCT00836381
Title: Assessment of Patient-reported Goal Attainment in the Treatment of Female Overactive Bladder (Phase Ⅳ)
Brief Title: Assessment of Patient-reported Goal Attainment in the Treatment of Female Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, KYU-SUNG LEE, Proffesor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-09-006
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Antimuscarinics; Patient-reported goal achievement
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolterodine ER (Experimental): Tolterodine ER 4mg once daily
  Interventions: Drug: Tolterodine extended-release (ER) 4mg
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolterodine extended-release (ER) 4mg — Tolterodine extended-release (ER) 4mg once daily for 12 weeks
  Other Names: Detrusitol ER 4mg
  Arms: Tolterodine ER
Drug: Placebo — Identical Placebo once daily
  Arms: Placebo

SUMMARY:
For many years, antimuscarinics have been first-line pharmacological treatment for OAB. A recent meta-analysis of randomised, controlled trials on antimuscarinic treatment of OAB concluded that the drugs provide significant improvements in OAB symptoms compared with placebo but that the benefits are of limited clinical significance. The analysis questioned the clinical significance of the trial results, one reason for which was the lack of data on the use of sensitive patient-driven criteria. Traditional symptomatic and urodynamic measures of treatment success may be meaningful to clinicians but often have little meaning to patients. Therefore, patient-reported outcomes (PROs), which provide a subjective measure of a patient's response to treatment, are useful. Recently, clinicians treating OAB have begun to recognize the value of PROs but still overlook the treatment efficacy in terms of patient-reported goal achievement (PGA).

Patients with OAB have combination of symptoms and the extent to which individual OAB symptoms affect patients varies. Also each patient can have different goal for the treatment. Therefore, assessing the degree of goal achievement in each patient can provide a new aspect of treatment benefit.

This controlled study will advance the understanding of OAB in terms of patient-centered treatments goals and goal achievement and will provide a new aspect of treatment benefit.

DETAILED DESCRIPTION:
1. Objectives

   1. Primary objective: To explore the "Patient-reported Goal Attainment (PGA)" after 12 weeks of treatment with tolterodine extended-release (ER) 4mg in female overactive bladder (OAB) patients.
   2. Secondary objective: To explore the patient-reported treatment goals and the efficacy of tolterodine on the patient-reported outcomes (PROs), micturition diary parameters, and safety parameters from baseline to 12 weeks of treatment in female OAB patients.
2. Specific aim

   : To compare the efficacy of tolterodine ER 4mg with that of placebo, on PROs in terms of PGA after 12 weeks of treatment in female OAB patients.
3. Experimental/research design

   1. 12-week randomized, placebo-controlled, double-blind, parallel-group, prospective study in Korean women with symptoms of OAB
   2. Treatment: Each patient will receive tolterodine ER (4 mg, qd) or placebo (randomized in the ratio of 1:1) for 12 weeks.
   3. Time schedule Start date: 01/Jan/2009 Finish date: 01/Sep/2009 Duration of washout: 7 days Duration of run-in: 7 days Duration of enrollment period: 5 months Duration of treatment period: 12 weeks Completion of analysis: 6 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Female aged ≥ 18 and ≤ 80 years
2. Symptoms of OAB as verified by the screening 3 day micturition diary, defined by:

   Mean urinary frequency ≥8 times/24 hours Mean number of urgency episodes ≥ 2 episode/24 hours
3. Symptoms of OAB for ≥ 3 months.
4. Ability and willingness to correctly complete the micturition diary and questionnaire
5. Capable of understanding and having signed the informed consent form after full discussion of the research nature of the treatment and its risks and benefits

Exclusion Criteria:

1. Subjects with stress incontinence or mixed stress/urge incontinence where stress incontinence is the predominant component based on prior history.
2. Significant hepatic or renal disease, defined as having twice the upper limit of the reference range for serum concentrations of aspartate amino- transferase (AST [SGOT]), alanine aminotransferase (ALT [SGPT]), alkaline phosphatase or creatinine.
3. Any condition that is a contraindication for anticholinergic treatment, including uncontrolled narrow-angled glaucoma, urinary retention or gastric retention
4. Symptomatic acute urinary tract infection (UTI) during the run-in period
5. Recurrent UTI defined as having been treated for symptomatic UTI > 4 times in the last year
6. Diagnosed or suspected interstitial cystitis
7. Clinically significant bladder outlet obstruction or poor detrusor function defined by clinical symptoms and investigator's opinion according to local standard of care
8. Previous history of major urethral and/or bladder surgery
9. History of radiation treatment (external or interstitial) to pelvic organs or external genitalia for any reason.
10. Subjects with neuropathology that could affect the lower urinary tract or nerve supply
11. Patients with marked cystocele or other clinically significant pelvic prolapse.
12. Subjects with current (within 2 years) urogenital neoplasms or malignancies including bladder, uterine or cervical cancer
13. Treatment within the 14 days preceding randomization, or expected to initiate treatment during the study with: Any anticholinergic drugs other than trial drug Any drug treatment for overactive bladder
14. On an unstable dosage of any drug with anticholinergic side effects, or expected to start such treatment during the study
15. Subjects currently taking tricyclic antidepressants, diuretics or alpha blockers who have not been on a stable dose of these medications for at least one month
16. Current administration of a selective serotonin reuptake inhibitor (SSRI) and has not been on a stable dose for at least three months
17. Receipt of any electrostimulation or bladder training within the 14 days before randomization, or expected to start such treatment during the study
18. An indwelling catheter or practicing intermittent self-catheterization
19. Use of any investigational drug within 1 months preceding the start of the study
20. Patients with chronic constipation or history of severe constipation
21. Pregnant or nursing women
22. Sexually active females of childbearing potential not using reliable contraception for at least 1 month prior to study start and not agreeing to use such methods during the entire study period and for at least 1 month thereafter *Reliable contraceptive methods are defined as intrauterine devices (IUDs), combination type contraceptive pills, hormonal implants, double barrier method, injectable contraceptives and surgical procedures (tubal ligation or vasectomy).
23. Any other condition which makes the patient unsuitable for inclusion.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Percentage of goal attainment using visual analog scale (VAS) at visit 3 and 4 | visit 3 (treatment 4 weeks) and 4 (treatment 12 weeks)

SECONDARY OUTCOMES:
Assessment of patient-reported treatment goal | visit 3 (treatment 4 weeks) and 4 (treatment 12 weeks)
Patient-reported outcomes | visit 3 (treatment 4 weeks) and 4 (treatment 12 weeks),
Micturition diary efficacy parameters | visit 3 (treatment 4 weeks) and 4 (treatment 12 weeks),
Safety parameters | visit 3 (treatment 4 weeks) and 4 (treatment 12 weeks),

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea